CLINICAL TRIAL: NCT01415713
Title: Phase I/II Trial of Biweekly S-1, Leucovorin, Oxaliplatin and Gemcitabine (SLOG) in Metastatic Pancreatic Adenocarcinoma
Brief Title: The Study of Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1211
Record Dates: First submitted 2011-07-06; First posted 2011-08-12 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: enroll the 80 patients in this trial
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Statin dose titration (Experimental): SLOG regimen:
  S-1 20-40 mg/m2/b.i.d., day 1-7;Leucovorin 20 mg/m2/b.i.d., day 1-7;Oxaliplatin 85 mg/m2 in 250 mL of D5W,given as 2-hour intra-venous infusion, day 1;Gemcitabine 800 mg/m2 in 250 mL of normal saline, given as fixed dose-rate infusion,day 1;After the administration of gemcitabine, the infusion line should be flushed with 20 ml of normal saline and then 50 ml of 5% glucose solution before the administration of oxaliplatin; Every 14 days, as one cycle.Prophylactic G-CSF or GM-CSF will not be allowed in this study. In case of grade 4 or complication neutropenia, patients may receive G-CSF according to the regulation of National Insurance Bureru treated with appropriate antibiotics. Therapeutic G-CSF may be used at the discretion of attending physicians.
  Interventions: Drug: S-1,Leucovorin,Oxaliplatin,Gemcitabine

INTERVENTIONS:
Drug: S-1,Leucovorin,Oxaliplatin,Gemcitabine — Biweekly S-1, Leucovorin, Oxaliplatin and Gemcitabine (SLOG) in metastatic pancreatic adenocarcinoma
  Other Names: G-CSF

SUMMARY:
Phase I part, Primary objective: the maximum tolerated dose of S-1 in the SLOG regimen Secondary objectives: the dose-limiting toxicity of the regimen Phase II part, Primary objective: Overall tumor response rate (by RECIST criteria) Secondary objectives: Disease control rate (Objective response rate (ORR) + stable disease ≧ 16 weeks), Time to tumor progression, Progression-free survival, Overall survival ,Safety profile, Biomarker study

DETAILED DESCRIPTION:
Phase I: 2~24 patients Phase II: Considering a design with p0 = 0.25 and p1 = 0.40 for which error is 0.10 and errors is 0.20, these constraints can be met with a two-stage Simon's design of 25 patients in the first stage and 27 patients in the second stage.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have cyto-/histologically confirmed, recurrent or metastatic adenocarcinoma of the pancreas (mPAC).
2. Patients must have no history of prior chemotherapy.
3. Patients with prior radiotherapy.
4. Patients' baseline ECOG performance status must be 2.
5. Patients' life expectancy must be 12 weeks or greater.
6. Patients' age must be 20 and 75.
7. Patients must have adequate bone marrow function.
8. Patients must have adequate liver and renal function.
9. All patients must be sign and give written informed consent.

Exclusion criteria:

1. Patients who have major abdominal surgery, radiotherapy.
2. Patients with central nervous system metastasis.
3. Patients with active infection.
4. Pregnant or breast-nursing women.
5. Patients with active cardiopulmonary disease.
6. Patients who have peripheral neuropathy > Grade I.
7. Patients who have serious concomitant systemic disorders.
8. Patients who have other prior or concurrent malignancy.
9. Patients who are under biologic treatment for their malignancy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
to determine the following items in patients with metastatic pancreatic adenocarcinoma receiving SLOG | one year
  Patients will be entered in cohorts of three. In any dose level of S-1, if none develops DLT as listed after the first two doses of SLOG chemotherapy, another cohort of 3 patients will be accrued to the next dose level. If at any time two or more patients develop DLT at the same dose level, the dose escalation will be terminated, and the prior dosage level will be considered the MTD.

SECONDARY OUTCOMES:
to evaluate the following items in patients with metastatic pancreatic adenocarcinoma receiving SLOG treatment, | one year
  9.2.1 Simon's optimal two-stage design will be used to determine the target patient number for the phase II part of this study. Using the approach, we test a null hypothesis that the true-response probability is less than an uninteresting level (p0) of 25% against the alternative hypothesis that the true response probability is at least as great as a target level (p1) of 40%. Response probabilities less than 25% will be considered inactive while response probabilities greater than 40% will be called highly effective.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph.D., Study Chair — National Institute of Cancer Research; Kelvin Kun-Chih Tsai, Ph.D., Principal Investigator — National Institute of Cancer Research
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiang NJ, Tsai KK, Hsiao CF, Yang SH, Hsiao HH, Shen WC, Hsu C, Lin YL, Chen JS, Shan YS, Chen LT. A multicenter, phase I/II trial of biweekly S-1, leucovorin, oxaliplatin and gemcitabine in metastatic pancreatic adenocarcinoma-TCOG T1211 study. Eur J Cancer. 2020 Jan;124:123-130. doi: 10.1016/j.ejca.2019.10.023. Epub 2019 Nov 22. PMID 31765987